CLINICAL TRIAL: NCT05061862
Title: Cardiac Implantable Electronic Device (CIED) Research Study
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: CIED Research Study
Record Dates: First submitted 2021-09-20; First posted 2021-09-30 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Arrhythmias, Cardiac; Bradycardia; Tachycardia
MeSH Terms: conditions — Arrhythmias, Cardiac; Bradycardia; Tachycardia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- CIED Indicated Subjects: Subjects indicated to receive a cardiac implantable electronic devices (CIEDs)
  Interventions: Device: cardiac implantable electronic devices (CIEDs)

INTERVENTIONS:
Device: cardiac implantable electronic devices (CIEDs) — Subjects will be implanted with various cardiac implantable electronic devices and followed according to their standard of care. Medical imaging will be collected at various stages of the implant procedure and/or non-invasive diagnostic collection at follow-up visits, as applicable.

SUMMARY:
The study is designed to collect data on Cardiovascular Implantable Electronic Device (CIED) information, implant procedure details, and/or patient characteristics to support development of future CIED products and procedures.

DETAILED DESCRIPTION:
This is a data collection, non-randomized, multi-center study. The study will consist of different cohorts with each cohort being independent from another cohort. Each cohort may have a distinct objective, cohort-specific subject population, procedures, and assessments. The study will follow subjects receiving routine care, who meet all of the inclusion criteria and none of the exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age.
2. Subject is willing and able to provide written informed consent.
3. Subject is willing and able to complete the study procedures and visits for the duration of data collection requirements

Exclusion Criteria:

1. Subject is unwilling or unable to comply with study procedures as defined in the protocol.
2. Subject with a medical condition that precludes the patient from participation in the opinion of the investigator.
3. Subject is enrolled in another study that could confound the results of this study, without documented pre-approval from a Medtronic study manager.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects who meet all inclusion criteria and none of the exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-03-06 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Product Development | 3 years
  Characterize Cardiovascular Implantable Electronic Device (CIED) information, implant procedure details and/or patient characteristics to support development of future CIED products and procedures.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (8):
  - The Cardiac & Vascular Institute, Gainesville, Florida
  - Georgia Arrhythmia Consultants, Macon, Georgia
  - Oregon Health & Science University Hospital, Portland, Oregon
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- UZ Leuven - Campus Gasthuisberg, Leuven, Belgium